CLINICAL TRIAL: NCT03078842
Title: Establishing the Optimal Dose of Therapeutic Zinc Supplementation for the Treatment of Acute Diarrhea in Under Five Children - a Dose Response Trial in a South Asian and a Sub-Saharan African Setting
Brief Title: Zinc Dosing Trial - Does Dose Reduction Reduce Side Effects But Retain Efficacy in Diarrhoea Management
Acronym: ZTDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayesha De Costa (Other)
Collaborators: Center for Public Health Kinetics (Other); Muhimbili University of Health and Allied Sciences (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Ayesha De Costa, Scientist, World Health Organization
Organization: World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC.0002738
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will get dispersible zinc tablets that, contain either 20 mg, 10 mg, or 5 mg of zinc. All tablets look and taste the same. Randomization and tablet package labelling was done in Geneva, and no-one at the trial sites knows the actual zinc content of tablets packaged for each participant number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zinc-20 (Active Comparator): Zinc tablets, 20 mg per day
  Interventions: Dietary Supplement: Zinc tablets, 20 mg per day
- Zinc-10 (Experimental): Zinc tablets, 10 mg per day
  Interventions: Dietary Supplement: Zinc tablets, 10 mg per day
- Zinc-05 (Experimental): Zinc tablets, 5 mg per day
  Interventions: Dietary Supplement: Zinc tablets, 5 mg per day

INTERVENTIONS:
Dietary Supplement: Zinc tablets, 20 mg per day — Participants will receive rehydration, dietary counseling, and 1 tablet per day for 14 days of zinc-tablets, each of which contains 20 mg of zinc
  Arms: Zinc-20
Dietary Supplement: Zinc tablets, 10 mg per day — Participants will receive rehydration, dietary counseling, and 1 tablet per day for 14 days of zinc-tablets, each of which contains 10 mg of zinc
  Arms: Zinc-10
Dietary Supplement: Zinc tablets, 5 mg per day — Participants will receive rehydration, dietary counseling, and 1 tablet per day for 14 days of zinc-tablets, each of which contains 5 mg of zinc
  Arms: Zinc-05

SUMMARY:
Diarrhoea continues to be a major cause of child deaths. Current treatment of acute watery diarrhoea includes oral rehydration solution (ORS), zinc and continued feeding. The use of zinc is based on a number of studies that showed that zinc reduces the duration and severity of diarrhoea. The recommended dose of zinc in 6-59 month old children is 20mg/day for 10-14 days. This dose is associated with an increased risk of vomiting. No dosing studies are available to determine the optimal dose of zinc, which while maintaining the benefits also has a low risk of vomiting.

The investigators will conduct a double-blind randomized controlled trial of three doses of zinc (20mg/day, 10mg/day and 5mg/day) in two settings - one in Sub-Saharan Africa and the other in South Asia. The study population will be 4500 children with diarrhoea of less than 72 hours duration who are aged 6-59 months. They will be recruited from outpatient health facilities. All enrolled children will receive ORS and continued feeding as recommended by the World Health Organization. Those allocated to the standard zinc dose will receive an oral dispersible tablet with 20mg zinc daily for 14 days. Those allocated to lower dose zinc will receive identical tablets with either 10mg or 5mg zinc daily for 14 days. Enrolled children will be followed by until recovery from diarrhoea or 15 days after enrolment, whichever is later. In addition, study children will be assessed again at thirty (30), forty-five (45), and sixty (60) days to estimate impact on post illness outcomes. Primary outcomes will be mean duration of diarrhoea, proportion of episodes that last longer than 5 days, mean number of stools and proportion of children with vomiting.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 59 completed months of age
* Acute diarrhoea of less than 3 days at the time of screening or dysentery, defined as visible blood in the stool, of less than 3 days at the time of screening
* Likely to stay within the study area for the next 2 months
* Written informed consent from caretaker

Exclusion Criteria:

* Presence of severe acute malnutrition (WHZ<-3 or oedema)
* Presence of severe dehydration that cannot be corrected in 4 to 6 hours
* Signs of severe pneumonia (WHO definition of pneumonia with danger signs), sepsis, rapid diagnostic test (RDT) -confirmed malaria or other severe illness
* Previously or currently enrolled in the study
* Currently enrolled in another study
* Other child currently enrolled in the study in the same household
* Not intending to remain in study area for the duration of the study
* Parents refuse participation in the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4500 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion with long duration of diarrhoea | Measured daily for 15 days
  Diarrhoea continuing beyond five days
Continuation of diarrhoea symptoms | Measured daily for 15 days
  Total number of loose or watery stools after enrolment
Proportion of children vomiting after zinc treatment | Measured daily for 15 days
  Vomiting within 30 minutes of administration of zinc tablet

SECONDARY OUTCOMES:
Proportion of children experiencing serious adverse events (SAEs) | Measured until 60 days
  Serious adverse events (life-threatening or requiring hospitalization)
Proportion with intermediate duration of diarrhoea | Measured daily for 15 days
  Diarrhoea continuing beyond three days
Proportion of guardians with positive attitude towards treatment | Day 15
  The guardians will be asked if was easy to administer the treatment, if they think the child liked the treatment, if they saw any changes in the children after the treatment and if they would recommend this treatment to their friends' children.
Treatment adherence | Measured daily for 15 days
  Mean number of tablets consumed by the study child during the 14 day treatment period.
Mean serum plasma zinc concentration at Days 1, 3, 7, 15, 21 and 30 | Days 1, 3, 7, 15, 21 and 30
  Mean serum plasma zinc concentration at Days 1, 3, 7, 15, 21 and 30
Illness symptoms between day 15 and 60 after the treatment | Days 30, 45, 60
  2-week period prevalence and number of days with diarrhoea, fever, or respiratory symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Bahl, MBBS, Study Director — World Health Organization
Locations (2):
- Centre for Public Health Kinetics, New Delhi, India
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The exact mechanism of data sharing has not yet been decided among the researchers. But the study is funded by an Organization (Bill & Melinda Gates Foundation) that requires data sharing.

REFERENCES:
- [Derived] Kisenge R, Dhingra U, Rees CA, Liu E, Dutta A, Saikat D, Dhingra P, Somji S, Sudfeld C, Simon J, Ashorn P, Sazawal S, Duggan CP, Manji K. Risk factors for moderate acute malnutrition among children with acute diarrhoea in India and Tanzania: a secondary analysis of data from a randomized trial. BMC Pediatr. 2024 Jan 19;24(1):56. doi: 10.1186/s12887-024-04551-2. PMID 38238656
- [Derived] Dhingra U, Kisenge R, Sudfeld CR, Dhingra P, Somji S, Dutta A, Bakari M, Deb S, Devi P, Liu E, Chauhan A, Kumar J, Semwal OP, Aboud S, Bahl R, Ashorn P, Simon J, Duggan CP, Sazawal S, Manji K. Lower-Dose Zinc for Childhood Diarrhea - A Randomized, Multicenter Trial. N Engl J Med. 2020 Sep 24;383(13):1231-1241. doi: 10.1056/NEJMoa1915905. PMID 32966722
- [Derived] Somji SS, Dhingra P, Dhingra U, Dutta A, Devi P, Kumar J, Deb S, Semwal OP, Sazawal S, Manji K, Kisenge R, Bakari M, Aboud S, Liu E, Sudfeld C, Duggan CP, Ashorn P, Bahl R, Simon JL. Effect of dose reduction of supplemental zinc for childhood diarrhoea: study protocol for a double-masked, randomised controlled trial in India and Tanzania. BMJ Paediatr Open. 2019 Apr 24;3(1):e000460. doi: 10.1136/bmjpo-2019-000460. eCollection 2019. PMID 31206083